CLINICAL TRIAL: NCT01996930
Title: A Prospective, Randomised Controlled Trial to Determine the Safety and Efficacy of Steroid Impregnated Tape Compared to Standard Therapy With Silver Nitrate in the Treatment of Over-granulating Peritoneal Dialysis Catheter Exit Sites
Brief Title: Steroid Impregnated Tape in the Treatment of Over-granulating Peritoneal Dialysis Exit Sites
Acronym: STOP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr. Lukas Foggensteiner, Consultant Nephrologist, University Hospital Birmingham NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RRK 4249; 2013-003867-76 (EudraCT Number)
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Peritoneal Dialysis; Continuous Ambulatory Peritoneal Dialysis; End Stage Renal Failure; Chronic Renal Failure
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Silver Nitrate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Haelan tape (steroid impregnated tape) (Active Comparator): Haelan tape, medicated tape for cutaneous use, containing 4mcg Fludroxycortide per centimetre squared.
  Maximum daily dosage of 0.1mg = 25cm squared per day. Application = once daily and left in situ for 24 hours Maximum duration of treatment = 28 days
  Interventions: Drug: Haelan tape (steroid impregnated tape)
- Silver nitrate (Active Comparator): Avoca caustic applicator 95% w/w cutaneous stick Cautery with silver nitrate cutaneous stick undertaken twice weekly Maximum duration of treatment = 28 days
  Interventions: Drug: Silver Nitrate

INTERVENTIONS:
Drug: Haelan tape (steroid impregnated tape) — Medicated plaster applied daily. Max daily dose = 0.1mg (25cm squared per day)Maximum duration of treatment = 28 days
  Other Names: MA PL00551/0014
  Arms: Haelan tape (steroid impregnated tape)
Drug: Silver Nitrate — Cautery with silver nitrate cutaneous stick undertaken twice weekly for a maximum duration of treatment = 28 days
  Other Names: Avoca Caustic Applicator 95% w/w cutaneous stick; MA PL04286/0005
  Arms: Silver nitrate

SUMMARY:
Kidney failure is a devastating illness requiring treatment with dialysis or transplantation to preserve life. Individuals unable to have transplants are managed by peritoneal dialysis (PD)or haemodialysis (HD). PD involves the placement of a soft, flexible plastic tube (catheter) into the abdomen, allowing dialysis fluid to be drained in and out of the peritoneal cavity. This catheter exits from a hole in the abdomen and occasionally patients can have complications at this exit site. One possible complication is over-granulation. Over-granulation occurs as the wound attempts to heal and the skin around the exit site becomes red,'wet','bumpy' and stands 'proud' of the surrounding skin. An over-granulating exit site can lead to discomfort, pain, bleeding and harbour infection. More serious complications include dialysis failure, sepsis and death. There are several ways to treat over-granulation but there is limited research evidence to demonstrate which treatment is best. The study aims to compare current standard treatment which involves the application of silver nitrate by qualified nursing staff to chemically burn the tissue away, with an alternative treatment which involves the application of steroid impregnated tape to the area of over-granulating tissue by the patient themselves.

DETAILED DESCRIPTION:
This study will be a United Kingdom wide multi-centre trial. A minimum of 40 patients in each arm will be recruited. Subjects will be identified using a standardised exit site assessment tool by PD nurses in participating units during the routine care of their PD population. Any subject with an over-granulating exit site deemed to meet the agreed standard for treatment will be invited to participate.

Therapy will be administered for two weeks followed by an additional two weeks if clinically indicated. Treatment must be according to randomisation for the first 28 days. If after 14 days the over-granulation is worse than at day 0, then a medical decision to continue treatment may be taken. A further two weeks of the designated treatment may then be administered although this can be discontinued at any point if a satisfactory clinical response is observed.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been established on PD for > 3 months
* Subject has an over-granulating exit site judged to require treatment according to standard (appendix 1)
* If patient has exit site infection, they must currently be treated with antibiotics and the site must be clinically improving.
* Subject is > 18 years of age
* Subject is able to give informed consent

Exclusion Criteria:

* Subject has had peritonitis treated in the previous month
* Subject has been treated with silver nitrate or topical steroids in the previous 2 weeks
* Subject is receiving oral steroids
* Patient is unable to give informed consent
* Patient is participating in a clinical trial of an intervention relating to PD catheters.
* Subject is pregnant or unwilling to use an effective method of contraception during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-12; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Complete response rate in over-granulation severity | 14 days
  The primary research objective of this study is to assess the total response at 14 days to treatment with either steroid tape or silver nitrate therapy on the over-granulated tissue surrounding the PD exit site.
  Assessment is by two blinded independent investigators (patient and therapy administrators will not be blinded to the therapy received). At each of the study visits, a series of photographs will be taken according to a study specific standard operating procedure and the two assessors will score the exit sites from the photographic series. There is no standardised scoring system for over-granulating exit sites so a scale has been devised:
  Score 1: Complete response:complete disappearance of over-granulation Score 2: Partial response: reduction in size or an obvious reduction in intensity of over-granulation Score 3: No change, appearance identical to that of pre-treatment Score 4: Worse, increase in size or increased intensity of over-granulation

SECONDARY OUTCOMES:
Partial response rate of over-granulation to treatment | 14 days and 28 days
  Partial response rate of over-granulation to treatment by either silver nitrate or steroid impregnated tape will assessed by two blinded independent investigators (patient and therapy administrators will not be blinded to the therapy received). At each of the study visits, a series of photographs will be taken according to a study specific standard operating procedure and the two assessors will score the exit sites from the photographic series. There is no standardised scoring system for over-granulating exit sites so a scale has been devised:
  Score 1: Complete response:complete disappearance of over-granulation Score 2: Partial response: reduction in size or an obvious reduction in intensity of over-granulation Score 3: No change, appearance identical to that of pre-treatment Score 4: Worse, increase in size or increased intensity of over-granulation
Recurrence of over-granulation | at 28 days and 56 days
  Following treatment, what is the rate of recurrence of over-granulation tissue at Day 28 and Day 56 of the study. The local investigators will assess the exit site at protocol defined study visits using a standardised exit site assessment tool.
Exit site infection rate | within 28 days and 56 days
  Following treatment, what is the rate of exit site infections within 28 and 56 days (An exit site infection is defined as occurring when a clinician decides treatment with antibiotics is required)
Exit site swab results | Baseline (Day 0), Day 7, Day 14, Day 21, Day 28 and Day 56
  At defined time points the exit site will be swabbed by trained staff to detect the presence of micro-organisms
Patient reported pain, discomfort and satisfaction score | Baseline (Day 0), Day 7, Day 14, Day 21, Day 28 and Day 56
  The study will assess patient reported pain and discomfort as well as satisfaction in terms of convenience and ease of use, with the treatment they received to treat their over-granulation tissue, through completion of a short non-validated patient questionnaire.
Occurrence of redness, ulceration or infection using a standardised exit site assessment tool | Baseline (Day 0), Day 7, Day 14, Day 21, Day 28, Day 56
  The local investigators will assess the exit site at protocol defined study visits using a standardised exit site assessment tool.

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Foggensteiner, BM FRCP PhD, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (8):
- United Kingdom (8):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Royal Devon & Exeter NHS Foundation Trust, Exeter
  - Hull and East Yorkshire Hospitals NHS Trust, Hull
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Royal Liverpool & Broadgreen University Hospitals NHS Trust, Liverpool
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - University Hospital of North Staffordshire NHS Trust, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No